CLINICAL TRIAL: NCT03044847
Title: The Cohort Study for Chronic Obstructive Pulmonary Diseases (COPD) in China---- Observation of the Disease Outcome and Identification of Prognostic Biomarkers for the Disease Outcome
Brief Title: The Cohort Study for Chronic Obstructive Pulmonary Disease (COPD) in China
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Kewu Huang, Professor/M.D., Beijing Chao Yang Hospital
Other Study IDs: 2016YFC0901102; ESR-16-12485 (Other: China-Japan Friendship Hospital, Ministry of Health)
Record Dates: First submitted 2017-01-25; First posted 2017-02-07 (Estimated); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: whole blood and sputum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- COPD group: The post-bronchodilator FEV1/FVC ratio < 0.70 was used as definition of COPD, which was proposed by the Global Initiative for Chronic Obstructive Lung Disease
  Interventions: Other: COPD group
- GOLD 0 group: GOLD 0 is defined as having chronic respiratory symptoms and/or high risk factors, but without airflow (post-BD FEV1/FVC ≥ 0.7). Chronic respiratory symptoms is defined as chronic cough, phlegm production, chest tightness, short of breath, dyspnea, wheeze, ect. High risk factors is defined as cigarette smoking, passive smoking, occupational exposures, bio-fuels exposures ect.

INTERVENTIONS:
Other: COPD group — The treatments will be determined by their treating physicians and no additional investigational drugs will be applied to the patients included in this study.
  Groups: COPD group

SUMMARY:
The purpose of this study is to establish the large COPD cohort and biological database in China, aiming for precision medicine to optimize diagnosis and treatment choices and to monitor and improve clinical outcomes in this disease.

DETAILED DESCRIPTION:
This is a 5-year multi-center observational prospective longitudinal cohort study to to establish the large COPD cohort and biological database in China, including COPD subjects( n= 3000) and GOLD 0 subjects (n= 800).Sites Investigators will be respiratory physicians working in the respiratory department of our sites, which must be tier 2 or tier 3 hospitals in China, with the equipment and ability to conduct pulmonary function test, HRCT.Patients must meet all the inclusion criteria and none of the exclusion criteria.No additional investigational drugs will be applied to the patients. Full analysis set will be used for all analyses. Missing data will be analysed as it is. Statistical analysis will be conducted by epidemiology & statistics work group from Chinese Academy of Sciences, using SAS and SUDAAN software. An electronic data capture system will be used in this study. Paper-based questionnaire administration will also be used.Questionnaire variables will be checked before data entry.During the study, PI will be in charge of the monitoring of the whole procedure. Two working group will do the data cleaning and data analysing.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-75 years
* COPD group: baseline post-bronchodilator FEV1/FVC < 0.7
* GOLD 0 group: individuals with chronic respiratory symptoms and/or high risk factors
* Signed informed consent obtained prior to participations with the ability to comply with protocol and be available for study visits over 5 years

Exclusion Criteria:

* Acute exacerbation in the past 3 months
* Having other respiratory diseases with massive lung tissue destruction such as severe bronchiectasis and tuberculosis, etc
* The usual criteria of serious uncontrolled diseases
* thoracic or abdominal surgery in the last 3 months
* eye surgery in the last three months
* retinal detachment
* myocardial infarction in the last 3 months
* admission to hospital for any cardiac condition in the last month
* heart rate over 120 beats per minute
* antibacterial chemotherapy for tuberculosis
* pregnant or breast feeding

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tier 2 or tier 3 hospitals in China
Sampling Method: Probability Sample
Enrollment: 3800 (Estimated)
Dates: Start 2016-07; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
COPD-related mortality and all-cause mortality | 10 years
  COPD-related mortality and all-cause mortality

SECONDARY OUTCOMES:
COPD exacerbation rate per year | 10 years
  COPD exacerbation rate per year

CONTACTS AND LOCATIONS:
Overall Officials: Kewu Huang, M.D., Study Director — Beijing Chao Yang Hospital
Locations (1):
- Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
no plan to share IPD

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03044847/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/47/NCT03044847/ICF_001.pdf